CLINICAL TRIAL: NCT02081105
Title: Bedside Assessment of PEEP-induced Lung Recruitment by Using Digital Chest-X-ray in ARDS Patients. A Multicenter Prospective Study.
Brief Title: Validation of Digital Chest-X-ray (CXR) to Assess Lung Recruitment in ARDS
Acronym: RECRUTEX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study stopped because it was difficult to recruit the 130 expected patients
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2013.818
Record Dates: First submitted 2014-02-27; First posted 2014-03-07 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: ARDS,; PEEP,; lung recruitment,; lung recruitability,; Chest-X-Ray,; lung imaging,; Pressure/Volume (PV) curve,; compliance,; respiratory mechanics
MeSH Terms: conditions — Respiratory Distress Syndrome; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEEP 5 (Other): level of PEEP of 5 cm H2O randomly applied to the patient
  Interventions: Other: PEEP of 5 or 15 cm H2O
- PEEP 15 (Other): level of PEEP of 15 cm H2O randomly applied to the patient
  Interventions: Other: PEEP of 5 or 15 cm H2O

INTERVENTIONS:
Other: PEEP of 5 or 15 cm H2O — PEEP of 5 or 15 cm H2O set at the respirator and applied to the patient for 10 minutes. Then, measurements are made at each PEEP in the following order: arterial blood gas, CXR, pressure-volume curve.

SUMMARY:
Lung recruitability is essential for optimal Positive end-expiratory pressure (PEEP) selection in ARDS patients. It is defined as the potential for the non aerated or poorly aerated lung mass to become aerated due to the increase in airway pressure. PEEP contributes to lung recruitment mostly by maintaining some amount of the end-inspiratory recruitment at the end of expiration. PEEP also stabilizes patency of the small airways and minimizes the repeated opening and closing of them during the breathing cycle, which is implicated in a further lung inflammation. The gold-standard method for assessing lung recruitability is lung CT scan. For economic and feasibility this technique cannot be used in routine. Therefore, techniques that can be used at the bedside to measure lung recruitability are very well known. The measurement of recruited lung volume (Vrec) by using pressure-volume curve generated by the ventilator is another reference method to approach lung recruitment. It can be done at the bedside. Chest-X-Ray (CXR) is an interesting option as done in routine in this setting. Furthermore, it allows quantifying aeration thanks numerical image processing and a regional approach. In a preliminary one-center study we found a significant negative correlation between the amount of Vrec and the reduction in lung density measured by digital CXR between 5 and 15 cm H2O PEEP. In present study we would like to extend this previous result on a larger number of patients in a multicenter investigation.

ELIGIBILITY:
Inclusion Criteria:

* intubation and mechanical ventilation in the ICU
* Ramsay score 6 under sedation and analgesia
* ICU respirator implemented with pressure-volume curve device
* age equal to or greater than 18 years
* ARDS defined from the Berlin criteria
* absence of pneumothorax on the CXR before the study
* Absence of pleural effusion greater than 500 ml estimated from ultrasonography.
* no child-bearing woman
* written inform consent signed by the next of kin

Exclusion Criteria:

* Pneumothorax
* Pleural effusion greater than 500 ml estimated from ultrasonography
* Thoracic surgery in the last 3 months
* Contra-indication to CXR
* contra-indication to PEEP of 15 cm H2O
* contra-indication to PEEP of 15 or PEEP 15 mandated
* pressure-volume curve not feasible
* refusal to participate
* language barrier of the next of kin
* child-bearing woman
* person under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-02; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of CXR to detect lung recruitability | At day 1
  1 CXR and 1 pressure-volume curve wil be performed at each PEEP for a given patient Determination of regions of interest in the posterior intercostal spaces of each lung in which density is measured to assess the total lung density at each PEEP. Measurement of Vrec between each PEEP level. One point per patient. Correlation of Vrec to change in density over all the patients and Receiver Operating Characteristic (ROC) curve of change in density to detect Vrec greater than 150 ml.

SECONDARY OUTCOMES:
static compliance | At day 1
  Static compliance will be analysed at each PEEP. End-expiratory and end-inspiratory occlusion during the tidal breath to measure the effective static compliance at each PEEP. Change in static compliance between PEEP levels.
oxygenation | At day 1
  Oxygenation will be evaluated at each PEEP. Arterial blood gas measured at the end of each PEEP application for Oxygen Pressure in arterial blood (PaO2) and PaO2/ Inhaled Oxygen Fraction (FIO2) ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Hodane Yonis, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Réanimation Médicale, Hôpital Croix-Rousse, Hospices Civils de Lyon, Lyon, France